CLINICAL TRIAL: NCT04839094
Title: Dry Nasopharyngeal Swab Versus Transported in Viral Transport Media Rapid Antigen Test Comparison for the Detection of SARS-CoV-2: a Comparative Trial (RESTART).
Brief Title: Dry Versus Wet Nasopharyngeal Rapid Test for the Detection of COVID-19.
Acronym: RESTART
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antonios Kritikos, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: Q2059
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2 diagnosis; RT-PCR; rapid antigen testing; saliva; viral transport medium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rapid antigen testing versus RT-PCR — Sensitivity of rapid antigen testing and RT-PCR performed on nasopharyngeal swabs versus saliva samples in COVID-19 hospitalized patients.

SUMMARY:
Saliva sampling could serve as an alternative non-invasive sample for SARS-CoV-2 diagnosis while rapid antigen testing (RAT) might help to mitigate the shortage of reagents sporadically encountered with RT-PCR. Thus, in the RESTART study the investigators compare antigen and RT-PCR testing methods on nasopharyngeal (NP) swabs and salivary samples. The investigators conducted a prospective observational study among COVID-19 hospitalized patients between 10th December 2020 and 1st February 2021. Paired saliva and NP samples were investigated by RT-PCR (Cobas 6800, Roche-Switzerland) and by two rapid antigen tests: One Step Immunoassay Exdia® COVID-19 Ag (Precision Biosensor, Korea) and Standard Q® COVID-19 Rapid Antigen Test (Roche-Switzerland).

DETAILED DESCRIPTION:
In response to the growing SARS-CoV-2 pandemic and shortages of laboratory based rapid molecular testing capacity and reagents on a worldwide scale, multiple manufacturers have developed rapid testing kits to use out of laboratory settings. These simple kits are based either on detection of proteins from the SARS-CoV-2 virus on respiratory samples (e.g. nasopharyngeal or throat swabs), or detection, in blood or serum, of human antibodies generated in response to infection.

On 28 October 2020 the Swiss Federal Council decided that as of 2 November 2020, in addition to polymerase chain reaction (PCR) tests, which are considered the "Gold standard" for SARS-CoV-2 diagnosis, it would be possible to conduct nasopharyngeal rapid antigen tests all over Switzerland, also outside licensed laboratories. In a hospital care setting rapid tests are intended to help physicians on prompt clinical management of cases with COVID-19 compatible symptoms upon admission and facilitate patient triage and flow, notably in a period marked of transition to higher incidence rates and enormous pressure on health system. This strategy was subsequently adopted by the University Hospital of Lausanne as well.

Roche's SARS-CoV-2 Rapid Antigen Test (which is the actual test employed by our institution) is a rapid chromatographic immunoassay intended for the qualitative detection of a specific antigen of SARS-CoV-2 present in human nasopharynx. This test is performed using a nasopharyngeal swab collected from a patient with a result available after 10-15 minutes. While the manufacturer reports very good diagnostic performances of the test, literature shows high variability of sensitivity and specificity.Rapid antigen test's diagnostic performances can be high enough to detect cases with high viral load (i.e. pre-symptomatic and early symptomatic cases up to five days from symptom onset. Because of the intense but short-lived nature of SARS-CoV-2 shedding form the upper respiratory tract, the clinical use of rapid antigen testing requires great attention to the timing of infection because testing late in the course of infection will cause an apparently low clinical sensitivity. There is a significant decline of the viral load after 5-7 days of symptoms. In order to account for this possible drawback and compensate the loss of rapid antigen test's diagnostic performance on late infection, a confirmatory RT-PCR is systematically performed by the microbiology laboratory of Lausanne University Hospital. So as to avoid multiple sampling of the same patient and accelerate time-to-final-results, a single nasopharyngeal swab is performed on each patient and soaked on a viral transport medium. From this transport medium both tests are performed (rapid antigen test and RT-PCR). This procedure, introduces a pre-dilution step (in contrast to the usual rapid antigen testing procedure using a dry nasopharyngeal swab) but is in accordance to the specifications of the manufacturers' instructions. While current literature advocates against a significant decrease of tests' analytical performances due to this strategy, there is no strong consensus regarding the influence of transport medium on viral load stability and on test's analytical and clinical sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged above 18 years with confirmed SARS-CoV-2 infection by RT-PCR assay.
* Provide informed consent.

Exclusion Criteria:

* Patient's refusal to participate in the study.
* Patients with negative RT-PCR if already performed for patient's follow up as part of standard care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized patients with a confirmed SARS-CoV-2 infection will be screened for inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic assessment | On the day of inclusion
  Comparison of diagnostic performances (sensitivity, specificity, positive and negative predictive value) of the different strategies on patients hospitalised with a SARS-CoV-2 infection.

SECONDARY OUTCOMES:
Limit of detection determination. | On the day of inclusion
  - Define the limit of detection viral load and lowest dilution with the highest positivity rate of both strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided